CLINICAL TRIAL: NCT05996068
Title: Enhancing Trauma Resuscitation Through Arterial Line Integration: A Before-After Study
Brief Title: Arterial Line in Trauma Resuscitation
Acronym: ALTR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202210095DINC
Record Dates: First submitted 2023-08-03; First posted 2023-08-16 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-08

CONDITIONS: Major Trauma
Keywords: major trauma; arterial line; resuscitation
MeSH Terms: interventions — Vascular Access Devices

STUDY DESIGN:
Intervention Model Description: We use se before-after study type and only the after phase receive intervention. Before phase will retrospectively collect data from patient without arterial line intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trauma patients with arterial line insertion (Active Comparator): the after phase, actively recruited patients who are eligible for arterial line insertion
  Interventions: Device: arterial line
- trauma patients without arterial line insertion (No Intervention): the before phase, retrospectively data collection from the past

INTERVENTIONS:
Device: arterial line — insert arterial line for patients who meet major trauma criteria
  Arms: trauma patients with arterial line insertion

SUMMARY:
Accident-related deaths is the 7th leading cause of death in Taiwan, and most of them is due to trauma from falls and traffic accident. Among trauma patients, the common cause of death is from hemorrhagic shock. Thus, real-time and accurate blood pressure monitoring is important for trauma patients. Incorrect blood pressure monitoring can lead to adverse events like traumatic cardiac arrest and shock and can also delay the time for intervention (fluid resuscitation, blood transfusion and operation). The current practice of blood pressure monitoring in trauma patient is by non-invasive blood pressure monitoring, which may be incorrect and not timely. Patient's body type and peripheral perfusion can both influence the result of non-invasive blood pressure monitoring.

With continuous and correct blood pressure monitoring, the resuscitation team can give adequate and timely treatment. In some trauma centers, arterial line insertion in trauma patients is a daily practice, while the evidence is inadequate and the potential benefit in unknown.

The main purpose of this study is to investigate the application of arterial line insertion in trauma patients. The study design is a prospective before-after study to exam whether arterial line insertion in trauma patients can reduce adverse event rate like hypovolemic shock and improve patient's outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale (GCS) 13 or less
* SBP < 90 mmHg
* Respiratory rate < 10 or > 29 breaths/min
* Fall from height > 6 meters
* High-Risk Auto Crash: Partial or complete ejection, intrusion > 30 cm any site, Need for extrication for entrapped patient, Death in passenger compartment
* Rider separated from transport vehicle with significant impact
* Penetrating injuries to head, neck, torso, and proximal extremities
* Skull deformity, suspected skull fracture
* Chest wall instability, deformity, or suspected flail chest
* Suspected pelvic fracture
* Suspected fracture of two or more proximal long bones
* Amputation proximal to wrist or ankle
* Active bleeding requiring a tourniquet or wound packing with continuous pressure
* Burns in conjunction with trauma

Exclusion Criteria:

* Pregnancy
* Patient or family who are unable to obtain informed consent
* Known coagulopathy that is inappropriate for arterial line insertion
* Known peripheral arterial occlusion disease that is inappropriate for arterial line insertion
* traumatic cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
composite primary endpoint (including any hypotension, vasopressors usage, any cardiac arrest in ER, Shock index ) | during ER stay, up to 6 hours
  including any hypotension, vasopressors usage, any cardiac arrest in ER, Shock index (HR/SBP)>1

SECONDARY OUTCOMES:
prolong ICU admission | up to 7 days
  define as > 6 days of admission
30 days mortality rate | mortality within 30 days of trauma event
  mortality within 30 days of trauma event
volume of fluid administration | during ER stay, up to 6 hours
  any type of fluid administration
Area under curve (AUC) difference under different time measuring frequency | 1/3/5/10 minutes
  We will use continuous blood pressure data and apply different intervals (1, 3, 5, and 10 minutes) to create a plot, then smooth it to calculate the area under the curve (AUC).
units of red blood cell transfusion | during ER stay, up to 6 hours
  units of red blood cell transfusion
arterial blood pressure trajectory | during ER stay, up to 6 hours
  We will depict the arterial blood pressure trajectory for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan

REFERENCES:
- [Background] Teixeira PG, Inaba K, Hadjizacharia P, Brown C, Salim A, Rhee P, Browder T, Noguchi TT, Demetriades D. Preventable or potentially preventable mortality at a mature trauma center. J Trauma. 2007 Dec;63(6):1338-46; discussion 1346-7. doi: 10.1097/TA.0b013e31815078ae. PMID 18212658
- [Background] Klauber MR, Marshall LF, Luerssen TG, Frankowski R, Tabaddor K, Eisenberg HM. Determinants of head injury mortality: importance of the low risk patient. Neurosurgery. 1989 Jan;24(1):31-6. doi: 10.1227/00006123-198901000-00005. PMID 2927596
- [Background] Eisenberg HM, Gary HE Jr, Aldrich EF, Saydjari C, Turner B, Foulkes MA, Jane JA, Marmarou A, Marshall LF, Young HF. Initial CT findings in 753 patients with severe head injury. A report from the NIH Traumatic Coma Data Bank. J Neurosurg. 1990 Nov;73(5):688-98. doi: 10.3171/jns.1990.73.5.0688. PMID 2213158
- [Background] Tieu BH, Holcomb JB, Schreiber MA. Coagulopathy: its pathophysiology and treatment in the injured patient. World J Surg. 2007 May;31(5):1055-64. doi: 10.1007/s00268-006-0653-9. PMID 17426904
- [Background] Schreiber MA, Meier EN, Tisherman SA, Kerby JD, Newgard CD, Brasel K, Egan D, Witham W, Williams C, Daya M, Beeson J, McCully BH, Wheeler S, Kannas D, May S, McKnight B, Hoyt DB; ROC Investigators. A controlled resuscitation strategy is feasible and safe in hypotensive trauma patients: results of a prospective randomized pilot trial. J Trauma Acute Care Surg. 2015 Apr;78(4):687-95; discussion 695-7. doi: 10.1097/TA.0000000000000600. PMID 25807399
- [Background] Wijnberge M, van der Ster B, Vlaar APJ, Hollmann MW, Geerts BF, Veelo DP. The Effect of Intermittent versus Continuous Non-Invasive Blood Pressure Monitoring on the Detection of Intraoperative Hypotension, a Sub-Study. J Clin Med. 2022 Jul 14;11(14):4083. doi: 10.3390/jcm11144083. PMID 35887844